CLINICAL TRIAL: NCT05858593
Title: Positive Youth Development in the Metaverse - Development of a Virtual Reality Afterschool Program for Middle Childhood Youth
Brief Title: Positive Youth Development in the Metaverse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Sun Joo (Grace) Ahn, PHD, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00006669
Record Dates: First submitted 2023-04-19; First posted 2023-05-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Healthy Lifestyle; Childhood ALL; Behavior, Child
Keywords: virtual reality; positive youth development; afterschool program
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Child Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to which study condition they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): In the treatment group, the child will receive the VR-based curriculum in addition to receiving the devices to use for 8 weeks.
  Interventions: Behavioral: Virtual reality curriculum
- Control (Active Comparator): In the control group, the child will still receive the devices to use for 8 weeks, but will not have the VR-based curriculum.
  Interventions: Behavioral: No Virtual reality curriculum

INTERVENTIONS:
Behavioral: Virtual reality curriculum — Rather than rely on mere exposure to devices, participants in the treatment group will receive a curriculum that integrates the devices into traditional content delivered through the after school program.
  Arms: Treatment
Behavioral: No Virtual reality curriculum — Children will be able to use the same devices but will not have access to a curriculum that integrates the devices with traditional content delivered through the after school program.
  Arms: Control

SUMMARY:
This pilot study aims to leverage VR's capacity to easily replicate content and allow for multiple users to share the same space and engage in activities as if they're meeting in person. Integrating VR into afterschool programs will allow youth to receive more consistent programming content, even when they are unable to travel to the physical location for the in-person meetings.

DETAILED DESCRIPTION:
This pilot study aims to leverage VR's capacity to easily replicate content and allow for multiple users to share the same space and engage in activities as if they're meeting in person. Integrating VR into afterschool programs will allow youth to receive more consistent programming content, even when they are unable to travel to the physical location for the in-person meetings. It will also empower youth to engage with the afterschool program at their own pace by providing a safe space to learn and practice their socioemotional skills. Implemented at scale, these benefits of a VR-integrated afterschool program will be able to address the issues of health inequity head on by expanding access to high quality afterschool content without incurring high operating costs. The results from this pilot study will provide a critical foundation to apply for an extramurally funded clinical trial to demonstrate the efficacy of a VR-integrated afterschool program on youth mental wellbeing.

Aim 1: Determine feasibility of a VR-integrated afterschool program where youth can access the VR content on their own at home.

Aim 2: Test the hypothesis that complementing the in-person afterschool program with VR will increase a) engagement and b) socioemotional competencies in youth.

Aim 3: Test the hypothesis that youth will demonstrate better mental wellbeing when the in-person afterschool program is complemented with VR.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the Chess & Community program
* Between the ages of 9-17
* The parent/primary caregiver of these children

Exclusion Criteria:

* Children who are unable to wear a VR headset will not be recruited

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Self-regulation | One-time assessment post-treatment (at 8 weeks)
  Early Adolescent Temperament Questionnaire-Revised ( 1-Almost always untrue, 2-Usually untrue, 3-Sometimes true, sometimes untrue, 4-Usually true, 5-Almost always true)
Mental well-being | One-time assessment post-treatment (at 8 weeks)
  Strengths and Difficulties Questionnaire (Not true = 0, Somewhat true = 1, Certainly true = 2)

SECONDARY OUTCOMES:
Engagement | 8 weeks
  Number of hours of programming delivered for both in-person and VR

CONTACTS AND LOCATIONS:
Locations (1):
- Athens Chess & Community, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data used in published analyses will be made available upon request to other researchers with a verified scientific purpose, guarantee that they will store the data securely, not share the data further, not attempt to use the data to determine the identities of research participants, and reference the source of the data in any resulting publications. Intellectual property rights to all software applications and hardware products will be maintained by the University of Georgia.
Supporting Information: Analytic Code
Access Criteria: Verified scientific purpose, guarantee that they will store the data securely, not share the data further, not attempt to use the data to determine the identities of research participants, and reference the source of the data in any resulting publications